CLINICAL TRIAL: NCT05867576
Title: Randomised Controlled Trial of Acceptance and Commitment Therapy in Tuberous Sclerosis Complex
Brief Title: Acceptance and Commitment Therapy in Tuberous Sclerosis Complex
Acronym: ACT in TSC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: The Tuberous Sclerosis Association (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CH/2020/7042
Record Dates: First submitted 2021-05-21; First posted 2023-05-22 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Tuberous Sclerosis Complex; Acceptance and Commitment Therapy; Mental Health; Psychology; Paediatrics; Neurology; Remote therapy; TAND
MeSH Terms: conditions — Tuberous Sclerosis; Psychological Well-Being | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial of 6-12 sessions of ACT versus waitlist control. Waitlist control will involve a delay in the offer of ACT sessions for 12 weeks.
Masking Description: The study design is an unblinded, waitlist-controlled, randomised controlled trial (RCT). Randomisation will be conducted using established randomisation software RedCap. Researchers will not be blind to trial arm allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allocated to treatment (Active Comparator): Patients randomly allocated to this arm will receive treatment immediately. They will receive 6-12 sessions of ACT while patients allocated to the waitlist control arm do no receive any treatment.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Allocated to waitlist control (No Intervention): Patients randomly allocated to this arm will receive a delay in the treatment they receive. After a 12-week wait they will receive 6-12 sessions of ACT, while patients allocated to the immediate treatment arm receive no treatment for an equal duration.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Acceptance and commitment therapy (ACT) is an evidence-based psychological therapy that has been successfully used to improve physical and mental health among children and adults with chronic conditions. It is a "third wave" cognitive behavioural therapy that encourages openness to and awareness of the present moment in order to help participants maintain behaviours consistent with their life goals. ACT fosters engagement with, rather than avoidance of, painful experiences to move towards acceptance of unchangeable difficulties alongside building a rich and meaningful life despite the presence of ongoing difficulties. This gives ACT strong face validity for application to TCS patients where there can be permanent cognitive impairment and unavoidable ongoing physical symptoms and functional limitations.
  Arms: Allocated to treatment

SUMMARY:
The study will assess the acceptability and feasibility of a randomised controlled trial of 6-12 sessions of remotely-delivered Acceptance and Commitment Therapy (ACT) versus waitlist control. Waitlist control will involve a delay in the offer of ACT sessions for 12 weeks. Participants may access all services as usual in this time. Follow-up assessments will be conducted at 12-, 24 and 48 weeks post-randomisation to measure effectiveness.

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is a genetic disease caused by mutations in the tumour suppressor genes TSC1 and TSC2. The clinical hallmarks of the disease are the growth of benign tumours in various organs such as the brain, kidneys and skin. Seizures are present in around 60% of the population and neurodevelopmental problems such as attention deficit disorder and autism are common. Anxiety and depressive disorders are similarly linked and at the psychosocial level, there is increasing evidence of the effect of TSC on self-esteem, family functioning and peer relationships resulting in poorer quality of life. Despite these difficulties, no unique treatments, and almost no effective evidenced psychological treatments for TSC are available.

This trial aims to assess the feasibility and acceptability of Acceptance and Commitment Therapy (ACT) as a psychological treatment to improve quality of life among adolescents and young adults with TSC. ACT is a cognitive behavioural therapy that helps participants accept difficulties that they are unable to change. There is strong evidence for ACT's clinical effectiveness amongst patients with chronic diseases. The intervention will be delivered to participants aged 11-24 with TSC and sufficient cognitive and speech capabilities to take part. This will be delivered remotely via secure video-conferencing software. Our primary hypothesis is that ACT will be acceptable and feasible delivered remotely and may yield clinical improvements in health and quality of life.

The study will be a 12-week, waitlist controlled randomised clinical trial. Participants will be randomised to receive 12-weeks treatment either immediately or following a 12-week wait. The treatment will be ACT adapted for 11-24-year olds who have TSC. Treatment will involve 6 to 12 weekly sessions of ACT of up to one hour each in length. Clinical outcomes will be assessed unblinded at baseline, 12, 24 and 48 weeks from randomisation. As a feasibility and acceptability study a range of physical and mental health outcomes are assessed. All clinical outcomes focus on health, wellbeing and quality of life from baseline to 12 week (3-month) follow-up amongst those offered ACT immediately versus waitlist controls.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11 to 24 years.
* Diagnosis of Tuberous Sclerosis Complex.
* Sufficient understanding of English to engage with the intervention (spoken and written), as judged by the assessing clinician.
* Sufficient cognitive, sensory and speech capabilities to take part in the intervention.
* Participants (or their parents if under 16) give verbal or written informed consent to participate in the study.
* Participants give verbal or written assent if under 16.
* Receiving treatment over video-conferencing will be the default modality for delivery, so access to the internet is a requirement.

Exclusion Criteria:

* Previous structured behavioural intervention within last 6 months.
* Previous or current alcohol/substance dependence, psychosis, suicidality, or anorexia nervosa.
* Moderate or severe intellectual disability.
* Immediate risk to self or others.
* Parent or child not able to speak, read or write English.

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Treatment completion rate | Assessed at 3-month follow-up.
  The proportion of patients showing interest who then consent to the trial and complete the intervention.
Treatment completion rate | Assessed at 6-month follow-up
  The proportion of patients showing interest who then consent to the trial and complete the intervention.
Session attendance rate | Assessed at 3-month follow-up
  The session attendance rate compared to feasibility benchmarks.
Session attendance rate | Assessed at 6-month follow-up
  The session attendance rate compared to feasibility benchmarks.
The credibility/expectancy questionnaire | Assessed at baseline
  Assessing participant ratings of treatment credibility. Minimum score = 5; maximum score = 45. Higher scores indicate better outcome.
The credibility/expectancy questionnaire | Assessed at session 2
  Assessing participant ratings of treatment credibility. Minimum score = 5; maximum score = 45. Higher scores indicate better outcome.
The experience of service questionnaire | Assessed at 3-month follow-up
  A questionnaire used nationally in child and adolescent mental health services completed by patients and parents/carers (if under 16) to assess participants' experience of the intervention. An additional item has been added to the experience of service questionnaire to assess video-conferencing treatment satisfaction. Minimum score = 0; maximum score = 20. Higher scores indicate better outcome.
The experience of service questionnaire | Assessed at 6-month follow-up
  A questionnaire used nationally in child and adolescent mental health services completed by patients and parents/carers (if under 16) to assess participants' experience of the intervention. An additional item has been added to the experience of service questionnaire to assess video-conferencing treatment satisfaction. Minimum score = 0; maximum score = 20. Higher scores indicate better outcome.

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire II | Assessed at 3, 6 and 12-month follow-up.
  A brief 7-item self-report measure assessing psychological inflexibility, which is the central treatment target for ACT. Validated for use among patients aged 16 and over. Minimum score = 7; maximum score = 49. Higher scores indicate worse outcome.
Avoidance and Fusion Questionnaire for Youth 8-items | Assessed at 3, 6 and 12-month follow-up.
  A brief self-report measure of psychological inflexibility, for children (11 to 15 year old participants). Minimum score = 0; maximum score = 32. Higher scores indicate worse outcome.
World Health Organisation wellbeing index 5-items | Assessed at 3, 6 and 12-month follow-up.
  A brief self-reported assessment of wellbeing and mental health. Minimum score = 7 score; maximum = 49. Higher scores indicate worse outcome. Minimum score = 0; maximum score = 49. Higher scores indicate worse outcome.
Generalised Anxiety Disorder assessment 7-items | Assessed at 3, 6 and 12-month follow-up.
  A brief self-reported measure of generalised anxiety symptoms using 4-point Likert scales based on diagnostic criteria. Minimum score = 0; maximum score = 21. Higher scores indicate worse outcome.
Patient Health Questionnaire 9-items | Assessed at 3, 6 and 12-month follow-up.
  Assesses symptoms of depression using self-reported 4-point Likert scales based on diagnostic criteria for major depression. Minimum score = 0; maximum score = 27. Higher scores indicate worse outcome.
Client Service Receipt Inventory | Assessed at 3, 6 and 12-month follow-up.
  A research instrument developed to collect information on service receipt, service-related issues and income. In addition, the Client Service Receipt Inventory collects information on school attendance in the 3-months prior to assessment.
TAND - TSC Associated Neuropsychiatric Disorders | Assessed at 3, 6 and 12-month follow-up.
  Assesses behavioural, intellectual, learning and psychiatric impact of TSC.
Pediatric Quality of Life Inventory (PedsQL) | Assessed at 3, 6 and 12-month follow-up.
  A 23-item generic health status instrument with parent and child forms that assesses five domains of health (physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning) in children and adolescents
Experiential interviews | Assessed at 3- and 6-month follow-up
  Participant experiences of treatment as described in semi-structured qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Sam Amin, MBCHB MSc PhD, Principal Investigator — University Hospitals Bristol & Weston NHS Trust
Locations (1):
- University Hospitals Bristol and Weston NHS Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No